CLINICAL TRIAL: NCT05207124
Title: Survey of Sarcopenia and Osteopenia in Individuals With Cerebral Palsy and Examination of Influences After Botulinum Neurotoxin Type A Injection
Brief Title: Sarcopenia and Osteopenia in Individuals With Cerebral Palsy and Influences After Botulinum Neurotoxin Type A Injection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-BR-108-088
Record Dates: First submitted 2021-10-04; First posted 2022-01-26 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Botulinum toxin injection group: onabotulinumtoxinA

SUMMARY:
Botulinum neurotoxin type A (BoNT-A) intervention to control the hypertonia of muscles is one of the evidence-based managements for children with spastic cerebral palsy. However, BoNT-A injection in animal models to induce weakness had revealed some detrimental effects on muscular and skeletal systems. There are some objectives of this research. The first aim is to establish the baseline data of deficiencies in bone condition and muscle mass for individuals with cerebral palsy. To confirm the influences of intramuscular administration of Botox on muscular and bony health in this population is the other aim.

DETAILED DESCRIPTION:
Individuals with cerebral palsy is vulnerable to osteopenia and sarcopenia. Botulinum neurotoxin type A (BoNT-A) intervention to control the hypertonia of muscles is one of the evidence-based managements for children with spastic cerebral palsy. However, BoNT-A injection in animal models to induce weakness had revealed some detrimental effects on muscular and skeletal systems. There are some objectives of this research. The first aim is to establish the baseline data of deficiencies in bone condition and muscle mass for individuals with cerebral palsy. To confirm the influences of intramuscular administration of Botox on muscular and bony health in this population is the other aim.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of spastic CP (cerebral palsy)
2. moderate to severe spasticity over the limbs, Modified Ashworth Scale score≧2

Exclusion Criteria:

1. fixed contractures of the limbs
2. previous musculoskeletal surgery on the limbs
3. contraindications to botulinum toxin intervention

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: cerebral palsy is vulnerable for osteopenia and sarcopenia
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
DXA (dual-energy x-ray absorptiometry) | change from baseline at 24 weeks after botulinum neurotoxin type A injection
  dual-energy x-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No